CLINICAL TRIAL: NCT03184870
Title: A Phase 1b/2 Study of BMS-813160 in Combination With Chemotherapy or Nivolumab in Patients With Advanced Solid Tumors
Brief Title: A Study of BMS-813160 in Combination With Chemotherapy or Nivolumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV202-103; 2017-001725-40 (EudraCT Number)
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — BMS-813160; Nivolumab; 130-nm albumin-bound paclitaxel; Gemcitabine; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1 Arm A [First-line (1L) Colorectal]: BMS-813160 followed by BMS-813160 + FOLFIRI (Experimental): FOLFIRI: FOL (folinic acid [leucovorin]) F (fluorouracil [5-fluorouracil]) IRI (irinotecan [CAMPTOSAR])
  Interventions: Drug: BMS-813160; Drug: 5-fluorouracil (5-FU); Drug: Leucovorin; Drug: Irinotecan
- Part 1 Arm B [1L Pancreatic]: BMS-813160 followed by BMS-813160 + Gemcitabine/Nab-paclitaxel (Experimental)
  Interventions: Drug: BMS-813160; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part 1 Arm C [2L Pancreatic & 2/3L Colorectal MSS]: BMS-813160 followed by BMS-813160 + Nivolumab (Experimental): 2L: Second-line 2/3L: Second/third-line MSS: Microsatellite stable
  Interventions: Drug: BMS-813160; Biological: Nivolumab
- Part 2 Arm A Cohort 1a [2L Colorectal]: BMS-813160 + FOLFIRI (Experimental)
  Interventions: Drug: BMS-813160; Drug: 5-fluorouracil (5-FU); Drug: Leucovorin; Drug: Irinotecan
- Part 2 Arm A Cohort 1b [2L Colorectal]: BMS-813160 + FOLFIRI (Experimental)
  Interventions: Drug: BMS-813160; Drug: 5-fluorouracil (5-FU); Drug: Leucovorin; Drug: Irinotecan
- Part 2 Arm A Cohort 1c [2L Colorectal]: FOLFIRI (Experimental)
  Interventions: Drug: 5-fluorouracil (5-FU); Drug: Leucovorin; Drug: Irinotecan
- Part 2 Arm B Cohort 3a [1L Pancreatic]: BMS-813160 + Gemcitabine/Nab-paclitaxel (Experimental)
  Interventions: Drug: BMS-813160; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part 2 Arm B Cohort 3b [1L Pancreatic]: BMS-813160 + Nivolumab + Gemcitabine/Nab-paclitaxel (Experimental)
  Interventions: Drug: BMS-813160; Biological: Nivolumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part 2 Arm B Cohort 3c [1L Pancreatic]: Gemcitabine/Nab-paclitaxel (Experimental)
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part 2 Arm C Cohort 4 [2L Pancreatic]: BMS-813160 + Nivolumab (Experimental)
  Interventions: Drug: BMS-813160; Biological: Nivolumab
- Part 2 Arm C Cohort 5 [2/3L Colorectal MSS]: BMS-813160 + Nivolumab (Experimental)
  Interventions: Drug: BMS-813160; Biological: Nivolumab
- Part 2 Arm D Cohort 7 [2L Pancreatic]: BMS-813160 Monotherapy (Experimental)
  Interventions: Drug: BMS-813160
- Part 2 Arm D Cohort 8 [2/3L Colorectal MSS]: BMS-813160 Monotherapy (Experimental)
  Interventions: Drug: BMS-813160

INTERVENTIONS:
Drug: BMS-813160 — Specified dose on specified days
  Arms: Part 1 Arm A [First-line (1L) Colorectal]: BMS-813160 followed by BMS-813160 + FOLFIRI; Part 1 Arm B [1L Pancreatic]: BMS-813160 followed by BMS-813160 + Gemcitabine/Nab-paclitaxel; Part 1 Arm C [2L Pancreatic & 2/3L Colorectal MSS]: BMS-813160 followed by BMS-813160 + Nivolumab; Part 2 Arm A Cohort 1a [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1b [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm B Cohort 3a [1L Pancreatic]: BMS-813160 + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3b [1L Pancreatic]: BMS-813160 + Nivolumab + Gemcitabine/Nab-paclitaxel; Part 2 Arm C Cohort 4 [2L Pancreatic]: BMS-813160 + Nivolumab; Part 2 Arm C Cohort 5 [2/3L Colorectal MSS]: BMS-813160 + Nivolumab; Part 2 Arm D Cohort 7 [2L Pancreatic]: BMS-813160 Monotherapy; Part 2 Arm D Cohort 8 [2/3L Colorectal MSS]: BMS-813160 Monotherapy
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Part 1 Arm C [2L Pancreatic & 2/3L Colorectal MSS]: BMS-813160 followed by BMS-813160 + Nivolumab; Part 2 Arm B Cohort 3b [1L Pancreatic]: BMS-813160 + Nivolumab + Gemcitabine/Nab-paclitaxel; Part 2 Arm C Cohort 4 [2L Pancreatic]: BMS-813160 + Nivolumab; Part 2 Arm C Cohort 5 [2/3L Colorectal MSS]: BMS-813160 + Nivolumab
Drug: Nab-paclitaxel — Specified dose on specified days
  Arms: Part 1 Arm B [1L Pancreatic]: BMS-813160 followed by BMS-813160 + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3a [1L Pancreatic]: BMS-813160 + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3b [1L Pancreatic]: BMS-813160 + Nivolumab + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3c [1L Pancreatic]: Gemcitabine/Nab-paclitaxel
Drug: Gemcitabine — Specified dose on specified days
  Arms: Part 1 Arm B [1L Pancreatic]: BMS-813160 followed by BMS-813160 + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3a [1L Pancreatic]: BMS-813160 + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3b [1L Pancreatic]: BMS-813160 + Nivolumab + Gemcitabine/Nab-paclitaxel; Part 2 Arm B Cohort 3c [1L Pancreatic]: Gemcitabine/Nab-paclitaxel
Drug: 5-fluorouracil (5-FU) — Specified dose on specified days
  Arms: Part 1 Arm A [First-line (1L) Colorectal]: BMS-813160 followed by BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1a [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1b [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1c [2L Colorectal]: FOLFIRI
Drug: Leucovorin — Specified dose on specified days
  Arms: Part 1 Arm A [First-line (1L) Colorectal]: BMS-813160 followed by BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1a [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1b [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1c [2L Colorectal]: FOLFIRI
Drug: Irinotecan — Specified dose on specified days
  Arms: Part 1 Arm A [First-line (1L) Colorectal]: BMS-813160 followed by BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1a [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1b [2L Colorectal]: BMS-813160 + FOLFIRI; Part 2 Arm A Cohort 1c [2L Colorectal]: FOLFIRI

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, drug levels, drug effects, and preliminary efficacy of BMS-813160 alone or in combination with either chemotherapy or nivolumab or chemotherapy plus nivolumab in participants with metastatic colorectal and pancreatic cancers.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have metastatic colorectal or pancreatic cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Ability to swallow pills or capsules
* Required to undergo mandatory pre and on-treatment biopsies
* Adequate marrow function
* Adequate other organ functions
* Ability to comply with study visits, treatment, procedures, pharmacokinetic (PK) and pharmacodynamic (PD) sample collection, and required study follow-up

Exclusion Criteria:

* Histology other than adenocarcinoma (neuroendocrine or acinar cell)
* Suspected, known, or central nervous system (CNS) metastases (Imaging required only if participants are symptomatic)
* Active, known or suspected autoimmune disease
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity
* Prior treatment with cysteine-cysteine chemokine receptor 2 (CCR2) and/or cysteine-cysteine chemokine receptor 5 (CCR5) inhibitors, programmed death-1 receptor (PD-1), programmed death-ligand 1 [PD(L)-1] or cytotoxic T-lymphocyte antigen-4 (CTLA-4) antibodies
* History of allergy to study treatments or any of its components of the study arm that participant is enrolling

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (40):
- United States (28):
  - Local Institution - 0003, Birmingham, Alabama
  - Local Institution - 0026, Phoenix, Arizona
  - Local Institution - 0002, Los Angeles, California
  - Local Institution - 0025, Los Angeles, California
  - Local Institution - 0041, Orange, California
  - Local Institution - 0015, Aurora, Colorado
  - Local Institution - 0018, Washington D.C., District of Columbia
  - Local Institution - 0048, Brooksville, Florida
  - Local Institution - 0047, St. Petersburg, Florida
  - Local Institution - 0005, Baltimore, Maryland
  - Local Institution - 0033, Boston, Massachusetts
  - Local Institution - 0027, Rochester, Minnesota
  - Local Institution - 0039, Hattiesburg, Mississippi
  - Local Institution - 0023, St Louis, Missouri
  - Local Institution - 0004, Hackensack, New Jersey
  - Local Institution - 0017, New York, New York
  - Local Institution - 0024, Rochester, New York
  - Local Institution - 0046, Charlotte, North Carolina
  - Local Institution - 0044, Cleveland, Ohio
  - Local Institution - 0021, Cleveland, Ohio
  - Local Institution - 0037, Allentown, Pennsylvania
  - Local Institution - 0014, Philadelphia, Pennsylvania
  - Local Institution - 0020, Philadelphia, Pennsylvania
  - Local Institution - 0045, Charleston, South Carolina
  - Local Institution - 0034, Nashville, Tennessee
  - Local Institution - 0038, Nashville, Tennessee
  - Local Institution - 0016, Salt Lake City, Utah
  - Local Institution - 0042, Charlottesville, Virginia
- Local Institution - 0028, Clayton, Victoria, Australia
- Belgium (3):
  - Local Institution - 0050, Brussels
  - Local Institution - 0051, Edegem
  - Local Institution - 0049, Leuven
- Canada (3):
  - Local Institution - 0013, Edmonton, Alberta
  - Local Institution - 0012, Ottawa, Ontario
  - Local Institution - 0001, Toronto, Ontario
- Germany (2):
  - Local Institution - 0022, Dresden
  - Local Institution - 0007, Heidelberg
- Spain (3):
  - Local Institution - 0031, Barcelona
  - Local Institution - 0032, Madrid
  - Local Institution - 0030, Majadahonda - Madrid

REFERENCES:
- [Derived] Le DT, Folprecht G, Varghese AM, Gutierrez M, Noel M, Trikalinos NA, Chen E, Dayyani F, Davis SL, Ma WW, BasuMallick A, Garrido-Laguna I, Osawa M, O'Brien S, Novosiadly RD, Xu K, Greenawalt DM, Dutta S, Twyman Saint Victor C, Lenz HJ. Phase 1b/2 study of BMS-813160, a CCR2/5 dual antagonist, in combination with chemotherapy or nivolumab in patients with advanced pancreatic or colorectal cancer. J Immunother Cancer. 2026 Jan 22;14(1):e011284. doi: 10.1136/jitc-2024-011284. PMID 41571299
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two additional cohorts (Part 2-Arm D-Cohorts 7 and 8) with 300 mg BMS-813160 twice per day were planned according to a previous version of the protocol. However, these cohorts did not open for enrollment due to Cohort 4 being closed due to futility per Revised Protocol 06.
Groups:
- Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI: First-line treatment BMS-813160 300 mg twice a day in combination with FOLFIRI in participants with metastatic colorectal cancer
- Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI: First-line treatment BMS-813160 600 mg once a day in combination with FOLFIRI in participants with metastatic colorectal cancer
- Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB: First-line treatment BMS-813160 300 mg twice a day in combination with Gem/nab-paclitaxel (ABRAXANE) in participants with pancreatic cancer
- Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB: First-line treatment BMS-813160 600 mg once a day in combination with Gem/ nab-paclitaxel (ABRAXANE)
- Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO: Second- and third-line treatment BMS-813160 300mg twice a day in combination with nivolumab in participants with microsatellite stable colorectal cancer
- Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO: Second- and third-line treatment BMS-813160 600mg once a day in combination with nivolumab in participants with microsatellite stable colorectal cancer
- Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO: Second- and third-line treatment BMS-813160 300mg once a day in combination with nivolumab in participants with microsatellite stable colorectal cancer
- Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO: Second- and third-line treatment BMS-813160 150mg once a day in combination with nivolumab in participants with microsatellite stable colorectal cancer
- Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO; Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO: Second-line treatment BMS-813160 300mg twice per day in combination with nivolumab in participants with pancreatic cancer
- Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO: Second-line treatment BMS-813160 600mg once per day in combination with nivolumab in participants with pancreatic cancer
- Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI: Second-line treatment BMS-813160 300mg twice per day in combination with FOLFIRI in participants with colorectal cancer
- Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI: Second-line treatment BMS-813160 150mg once per day in combination with FOLFIRI in participants with colorectal cancer
- Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI: Second-line treatment FOLFIRI in participants with colorectal cancer.
  9 of the 26 participants who originated in this arm crossed over to Cohort 5.
- Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB: First-line treatment BMS-813160 300mg twice per day in combination with gemcitabine/nab-paclitaxel in participants with pancreatic cancer
- Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO: First-line treatment BMS-813160 300mg twice per day in combination with gemcitabine/nab-paclitaxel and nivolumab in participants with pancreatic cancer
- Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB: First-line treatment gemcitabine/ nab-paclitaxel in participants with pancreatic cancer
- Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO: Second- and third-line treatment BMS-813160 300mg twice per day in combination with nivolumab in participants with microsatellite stable colorectal cancer
Period: Initial Treatment
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Started | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 (9 of the original 26 participants in Cohort 1c were allowed to cross over to Cohort 5 if it was in their best interest as determined by their treating physician and participants meet all eligibility criteria.) | 35 | 35 | 32 | 24 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 24
Not completed — Death | 6 | 6 | 8 | 8 | 6 | 6 | 6 | 7 | 1 | 2 | 26 | 28 | 10 | 33 | 34 | 26 | 20 | 18
Not completed — Other Reasons | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 2 | 2 | 0 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 5 | 2 | 2
Not completed — Moved to crossover treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0
Period: Crossover Treatment
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Started (Participants who received crossover treatment) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 (9 of the original 26 participants in Cohort 1c were allowed to cross over to Cohort 5 if it was in their best interest as determined by their treating physician and participants meet all eligibility criteria.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO | Total
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33 | 324
Age, Continuous [Mean (Full Range); unit: Years] — Population: 9 participants crossed over from Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI to Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO. The baseline characteristics are broken into two rows to prevent double-counting and to make it the data associated with the cross over participants clear.
  Years
    All Cohorts except Part 2-Arm C-Cohort 5: number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 0 | 291
    All Cohorts except Part 2-Arm C-Cohort 5 | 65.6 [54 to 83] | 53.3 [28 to 66] | 64.1 [54 to 80] | 62.7 [51 to 80] | 59.5 [48 to 76] | 61.7 [52 to 66] | 45.1 [33 to 57] | 60.5 [42 to 77] | 61.0 [61 to 61] | 50.0 [49 to 51] | 55.0 [29 to 76] | 58.9 [30 to 83] | 57.9 [37 to 77] | 65.9 [46 to 76] | 65.3 [43 to 85] | 65.5 [49 to 84] | 63.9 [34 to 77] |  | 61.4 [28 to 85]
    Part 2-Arm C-Cohort 5 only: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 33
    Part 2-Arm C-Cohort 5 only |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 55.0 [39 to 69] | 55.0 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 9 participants crossed over from Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI to Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO. The baseline characteristics are broken into two rows to prevent double-counting and to make it the data associated with the cross over participants clear.
  Participants
    All Cohorts except Part 2-Arm C-Cohort 5: number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 0 | 291
    All Cohorts except Part 2-Arm C-Cohort 5: Female | 3 | 2 | 6 | 6 | 2 | 3 | 3 | 3 | 1 | 0 | 13 | 11 | 9 | 15 | 15 | 15 | 8 |  | 115
    All Cohorts except Part 2-Arm C-Cohort 5: Male | 7 | 6 | 4 | 5 | 6 | 4 | 4 | 8 | 0 | 2 | 19 | 21 | 17 | 20 | 20 | 17 | 16 |  | 176
    Part 2-Arm C-Cohort 5 only: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 33
    Part 2-Arm C-Cohort 5 only: Female |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 18 | 18
    Part 2-Arm C-Cohort 5 only: Male |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 15 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 9 participants crossed over from Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI to Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO. The baseline characteristics are broken into two rows to prevent double-counting and to make it the data associated with the cross over participants clear.
  Participants
    All Cohorts except Part 2-Arm C-Cohort 5: number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 0 | 291
    All Cohorts except Part 2-Arm C-Cohort 5: Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 7 | 2 | 2 | 2 | 1 | 4 | 0 |  | 23
    All Cohorts except Part 2-Arm C-Cohort 5: Not Hispanic or Latino | 8 | 5 | 8 | 9 | 8 | 7 | 6 | 7 | 0 | 2 | 21 | 26 | 17 | 28 | 30 | 24 | 21 |  | 227
    All Cohorts except Part 2-Arm C-Cohort 5: Unknown or Not Reported | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 4 | 7 | 5 | 4 | 4 | 3 |  | 41
    Part 2-Arm C-Cohort 5 only: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 33
    Part 2-Arm C-Cohort 5 only: Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4 | 4
    Part 2-Arm C-Cohort 5 only: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 23 | 23
    Part 2-Arm C-Cohort 5 only: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 9 participants crossed over from Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI to Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO. The baseline characteristics are broken into two rows to prevent double-counting and to make it the data associated with the cross over participants clear.
  Participants
    All Cohorts except Part 2-Arm C-Cohort 5: number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 0 | 291
    All Cohorts except Part 2-Arm C-Cohort 5: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
    All Cohorts except Part 2-Arm C-Cohort 5: Asian | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 1 | 1 |  | 17
    All Cohorts except Part 2-Arm C-Cohort 5: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
    All Cohorts except Part 2-Arm C-Cohort 5: Black or African American | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 0 |  | 10
    All Cohorts except Part 2-Arm C-Cohort 5: White | 8 | 4 | 10 | 11 | 8 | 5 | 7 | 7 | 1 | 2 | 28 | 26 | 22 | 32 | 34 | 27 | 22 |  | 254
    All Cohorts except Part 2-Arm C-Cohort 5: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
    All Cohorts except Part 2-Arm C-Cohort 5: Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1 |  | 10
    Part 2-Arm C-Cohort 5 only: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 33
    Part 2-Arm C-Cohort 5 only: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 | 0
    Part 2-Arm C-Cohort 5 only: Asian |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1 | 1
    Part 2-Arm C-Cohort 5 only: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 | 0
    Part 2-Arm C-Cohort 5 only: Black or African American |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3 | 3
    Part 2-Arm C-Cohort 5 only: White |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 28 | 28
    Part 2-Arm C-Cohort 5 only: More than one race |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0 | 0
    Part 2-Arm C-Cohort 5 only: Unknown or Not Reported |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days post last dose, up to approximately 3 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 25 | 35 | 35 | 31 | 23 | 32

2. Primary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose up to 100 days post last dose, up to approximately 3 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants | 5 | 5 | 5 | 7 | 5 | 6 | 6 | 6 | 1 | 2 | 12 | 12 | 6 | 24 | 22 | 15 | 17 | 19

3. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: Dose-limiting toxicities (DLTs) are severe adverse effects (AEs) that are attributed to BMS-813160 or the combination regimen and define the maximum tolerated dose of a medicine. DLTs will be defined based on the incidence, duration and grade of AEs for which no alternate cause can be identified. AEs will be evaluated according to the NCI CTCAE v4.03. The incidence of DLT(s) during the first 6 weeks of treatment in Part 1 (the DLT evaluation period) and 4 weeks for Part 2 will be used.
Time Frame: From first dose up to 100 days post last dose, up to approximately 3 years
Population: All treated participants who completed the DLT evaluation period
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: An Adverse Event (AE) leading to discontinuation is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment that leads to the discontinuation of study treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days post last dose, up to approximately 3 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants | 2 | 0 | 1 | 6 | 0 | 1 | 0 | 1 | 0 | 1 | 10 | 6 | 2 | 12 | 8 | 3 | 4 | 2

5. Primary Outcome: Number of Participants Who Died
Description: The number of participants who died within 100 days after receiving their last dose
Time Frame: From first dose up to 100 days post last dose, up to approximately 3 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants | 6 | 6 | 8 | 8 | 6 | 6 | 6 | 7 | 1 | 2 | 26 | 28 | 17 | 33 | 34 | 26 | 20 | 25

6. Primary Outcome: Number of Participants Experiencing Laboratory Abnormalities
Description: The number of participants experiencing laboratory abnormalities in pre-specified selected parameters during the treatment period per CTCAE (Version 4). Laboratory abnormalities are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days post last dose, up to approximately 3 years
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants
  ALANINE AMINOTRANSFERASE (ALT), LOCAL LAB (U/L) - Abnormal High: number analyzed (Participants) | 10 | 8 | 9 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 31 | 32 | 25 | 34 | 35 | 31 | 22 | 33
  ALANINE AMINOTRANSFERASE (ALT), LOCAL LAB (U/L) - Abnormal High | 2 | 4 | 5 | 7 | 2 | 1 | 3 | 6 | 1 | 1 | 15 | 9 | 10 | 24 | 28 | 24 | 10 | 13
  ASPARTATE AMINOTRANSFERASE (AST), LOCAL LAB (U/L) - Abnormal High: number analyzed (Participants) | 10 | 8 | 9 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 31 | 32 | 25 | 34 | 35 | 31 | 21 | 33
  ASPARTATE AMINOTRANSFERASE (AST), LOCAL LAB (U/L) - Abnormal High | 2 | 4 | 5 | 7 | 3 | 3 | 5 | 5 | 1 | 1 | 15 | 12 | 9 | 21 | 26 | 24 | 12 | 19
  Total Bilirubin (UMOL/L) - Abnormal High: number analyzed (Participants) | 10 | 8 | 9 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 31 | 32 | 25 | 34 | 35 | 31 | 22 | 33
  Total Bilirubin (UMOL/L) - Abnormal High | 2 | 4 | 5 | 2 | 1 | 1 | 4 | 3 | 1 | 1 | 5 | 5 | 2 | 8 | 7 | 5 | 6 | 7
  Neutrophils (Absolute) (10^9/L) - Abnormal Low: number analyzed (Participants) | 10 | 8 | 9 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 31 | 32 | 25 | 35 | 35 | 31 | 22 | 33
  Neutrophils (Absolute) (10^9/L) - Abnormal Low | 6 | 4 | 5 | 9 | 2 | 1 | 1 | 2 | 0 | 0 | 25 | 20 | 18 | 22 | 25 | 25 | 1 | 4
  PLATELET COUNT (10^9/L) - Abnormal Low: number analyzed (Participants) | 10 | 8 | 9 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 31 | 32 | 25 | 35 | 35 | 31 | 22 | 33
  PLATELET COUNT (10^9/L) - Abnormal Low | 5 | 1 | 5 | 5 | 2 | 1 | 1 | 3 | 0 | 0 | 11 | 15 | 8 | 24 | 28 | 26 | 10 | 5

7. Primary Outcome: Vital Signs
Description: Vital sign measurements at baseline and at the end of treatment. Baseline evaluations will be defined as evaluations with a date on or prior to the day of first dose of study treatment.
Time Frame: From first dose to 100 days post last dose, up to approximately 3 years
Population: All treated participants with vital sign measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 1 | 3 | 5 | 4 | 7 | 3 | 7 | 10 | 1 | 1 | 9 | 9 | 5 | 21 | 24 | 16 | 15 | 24
mmHg
  Systolic Blood Pressure (mmHg) - End of Treatment: number analyzed (Participants) | 1 | 3 | 5 | 4 | 7 | 3 | 7 | 10 | 1 | 1 | 3 | 2 | 1 | 21 | 24 | 16 | 15 | 24
  Systolic Blood Pressure (mmHg) - End of Treatment | 133.0 (NA) — Standard deviation not calculated due to insufficient number of events | 129.7 (6.7) | 130.2 (21.8) | 143.0 (34.0) | 114.0 (15.0) | 125.0 (6.1) | 140.3 (18.0) | 124.0 (23.7) | 151.0 (NA) — Standard deviation not calculated due to insufficient number of events | 107.0 (NA) — Standard deviation not calculated due to insufficient number of events | 126.0 (15.9) | 113.0 (NA) — Standard deviation not calculated due to insufficient number of events | 113.0 (NA) — Standard deviation not calculated due to insufficient number of events | 123.2 (18.8) | 128.9 (17.8) | 118.8 (15.9) | 112.6 (11.6) | 123.1 (13.6)
  Systolic Blood Pressure (mmHg) - Follow-up: number analyzed (Participants) | 1 | 2 | 1 | 4 | 2 | 1 | 1 | 2 | 0 | 0 | 9 | 9 | 5 | 5 | 5 | 3 | 1 | 2
  Systolic Blood Pressure (mmHg) - Follow-up | 140.0 (8.5) | 124.5 (2.1) | 100.0 (NA) — Standard deviation not calculated due to insufficient number of events | 143.0 (34.0) | 140.0 (8.5) | 108.0 (NA) — Standard deviation not calculated due to insufficient number of events | 148.0 (NA) — Standard deviation not calculated due to insufficient number of events | 129.5 (29.0) |  |  | 127.9 (13.2) | 131.3 (20.6) | 113.6 (8.1) | 119.2 (15.1) | 142.6 (16.0) | 108.3 (30.1) | 113.0 (NA) — Standard deviation not calculated due to insufficient number of events | 113.5 (6.4)
  Diastolic Blood Pressure (mmHg) - End of Treatment: number analyzed (Participants) | 1 | 3 | 5 | 4 | 7 | 3 | 7 | 10 | 1 | 1 | 3 | 2 | 1 | 21 | 24 | 16 | 15 | 24
  Diastolic Blood Pressure (mmHg) - End of Treatment | 83.0 (NA) — Standard deviation not calculated due to insufficient number of events | 73.3 (7.2) | 75.4 (12.4) | 80.8 (17.7) | 69.6 (9.4) | 86.0 (18.2) | 89.7 (11.1) | 74.3 (11.3) | 86.0 (NA) — Standard deviation not calculated due to insufficient number of events | 67.0 (NA) — Standard deviation not calculated due to insufficient number of events | 79.0 (11.5) | 74.5 (3.5) | 75.0 (NA) — Standard deviation not calculated due to insufficient number of events | 69.2 (8.2) | 74.3 (8.6) | 70.2 (8.6) | 68.1 (6.5) | 74.3 (9.7)
  Diastolic Blood Pressure (mmHg)- Follow-up: number analyzed (Participants) | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 9 | 9 | 5 | 5 | 5 | 3 | 1 | 2
  Diastolic Blood Pressure (mmHg)- Follow-up | 79.0 (NA) — Standard deviation not calculated due to insufficient number of events | 71.5 (14.8) | 59.0 (NA) — Standard deviation not calculated due to insufficient number of events |  | 85.0 (2.8) | 69.0 (NA) — Standard deviation not calculated due to insufficient number of events | 98.0 (NA) — Standard deviation not calculated due to insufficient number of events | 72.5 (4.9) |  |  | 76.6 (14.6) | 76.1 (11.0) | 78.2 (7.3) | 68.0 (9.9) | 70.2 (10.5) | 66.7 (20.1) | 85.0 (NA) — Standard deviation not calculated due to insufficient number of events | 69.0 (2.8)

8. Primary Outcome: Number of Participants With Out-of-Range Electrocardiograms (ECG)
Description: The number of participants with ECG measurements outside of the range pre-specified in the protocol.
Time Frame: From baseline up to 100 days post last dose
Population: All treated participants with out-of-range ECGs
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 10 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 31 | 25 | 34 | 34 | 29 | 24 | 33
Participants
  QTcF INTERVAL (MSEC) < 450 | 7 | 8 | 10 | 8 | 8 | 7 | 7 | 10 | 1 | 2 | 31 | 27 | 23 | 26 | 30 | 26 | 24 | 31
  QTcF INTERVAL (MSEC): 450 <= QTcF < 480 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 6 | 4 | 3 | 0 | 2
  480<=QTcF<500 (MSEC) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  QTcF>= 500 (MSEC) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  QTcB INTERVAL (MSEC) < 450 | 4 | 7 | 8 | 5 | 7 | 3 | 3 | 7 | 1 | 2 | 20 | 21 | 15 | 14 | 17 | 19 | 21 | 15
  450<=QTcB<480 (MSEC) | 5 | 1 | 1 | 3 | 1 | 4 | 3 | 2 | 0 | 0 | 11 | 7 | 10 | 14 | 14 | 8 | 3 | 18
  480<=QTcB<500 (MSEC) | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3 | 0 | 4 | 3 | 2 | 0 | 0
  QTcB>= 500 (MSEC) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0

9. Primary Outcome: Percent Change in Regulatory T Cells (Treg) in Tumor Samples
Description: The percent change in Regulatory T Cells (Treg) were taken at prespecified timepoints. Baseline is defined as the last non-missing value prior to the first dosing.
Time Frame: From first dose up to prespecified timepoints listed below (C0D7; C0D14; C1D1; C1D15; C1D16; C1D28; C2D1)
Population: All treated participants with immunohistochemistry data
Measure: Median (Full Range); unit: Percent change in Treg
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 5 | 5 | 4 | 6 | 0 | 1 | 6 | 3 | 5 | 5 | 6 | 3 | 4 | 5
Percent change in Treg
  FOXP3 - C0D7: number analyzed (Participants) | 6 | 4 | 3 | 3 | 5 | 2 | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FOXP3 - C0D7 | 26.6 [-67 to 180] | -43.8 [-58 to -15] | -22.9 [-74 to -14] | 156.4 [-12 to 177] | 57.3 [-76 to 116] | -18.4 [-27 to -9] | -92.2 [-94 to 27] | 96.4 [14 to 152] |  | 101.0 [101 to 101] |  |  |  |  |  |  |  |
  FOXP3 - C0D14: number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 5 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FOXP3 - C0D14 | 26.5 [-50 to 103] | -19.8 [-78 to 53] | 60.0 [60 to 60] | -41.6 [-67 to -16] | -41 [-41 to -41] | -26.5 [-57 to 249] | 180.2 [-60 to 421] | -3.7 [-9 to 25] |  |  |  |  |  |  |  |  |  |
  FOXP3 - C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FOXP3 - C1D1 |  |  |  |  | 34.7 [-58 to 128] | 49 [49 to 49] | 147.4 [20 to 275] | 33.0 [-51 to 338] |  | 31.0 [31 to 31] |  |  |  |  |  |  |  |
  FOXP3 - C1D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 1 | 0
  FOXP3 - C1D15 |  |  |  |  | -25.9 [-48 to -6] | 14.5 [-90 to 322] | 39.1 [4 to 74] | -33 [-33 to -33] |  |  |  | -39.1 [-46 to -32] | 60 [60 to 60] | 113.6 [-1 to 228] |  | 17.0 [-39 to 73] | -64 [-64 to -64] |
  FOXP3 - C1D16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  FOXP3 - C1D16 |  |  |  |  |  |  |  |  |  |  | -21 [-21 to -21] |  |  |  |  |  |  |
  FOXP3 - C1D28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 5 | 5 | 6 | 3 | 4 | 5
  FOXP3 - C1D28 |  |  |  |  |  |  |  |  |  |  | -7.4 [-26 to 113] | -77.0 [-93 to -61] | 12.0 [-73 to 152] | -36.0 [-77 to -5] | 99.4 [-96 to 2199] | -46.6 [-55 to 551] | 216.7 [98 to 363] | -13.6 [-78 to 149]
  FOXP3 - C2D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  FOXP3 - C2D1 |  |  |  |  |  |  |  |  |  |  | 305.2 [-73 to 683] |  |  |  |  | 184 [184 to 184] | -2.4 [-37 to 32] | 156.2 [13 to 299]

10. Primary Outcome: Percent Change in Tumor-Associated Macrophages (TAMs) in Tumor Samples
Description: The percent change in Tumor-Associated Macrophages (TAMs) were taken at prespecified timepoints. Baseline is defined as the last non-missing value prior to the first dosing.
Time Frame: From first dose up to prespecified timepoints listed below (C0D7; C0D14; C1D1; C1D15; C1D16; C1D28; C2D1)
Population: All treated participants with immunohistochemistry data
Measure: Median (Full Range); unit: Percent change in TAM
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 0 | 0 | 6 | 3 | 4 | 5 | 6 | 3 | 0 | 2
Percent change in TAM
  CD163 Positive - C0D7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD163 Positive - C0D7 |  |  |  |  |  |  | 13.1 [2 to 808] | -12.7 [-67 to 231] |  |  |  |  |  |  |  |  |  |
  CD163 Positive - C0D14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD163 Positive - C0D14 |  |  |  |  |  |  | 95.4 [34 to 157] | 133.6 [0 to 286] |  |  |  |  |  |  |  |  |  |
  CD163 Positive - C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD163 Positive - C1D1 |  |  |  |  |  |  | 477.5 [334 to 621] | 22.1 [-28 to 520] |  |  |  |  |  |  |  |  |  |
  CD163 Positive - C1D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 2 | 0 | 0
  CD163 Positive - C1D15 |  |  |  |  |  |  | 7.6 [-37 to 53] | -93 [-93 to -93] |  |  |  | 89.8 [35 to 132] | -61 [-61 to -61] | 145.7 [43 to 248] |  | 60.3 [1 to 120] |  |
  CD163 Positive - C1D16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD163 Positive - C1D16 |  |  |  |  |  |  |  |  |  |  | 1369 [1369 to 1369] |  |  |  |  |  |  |
  CD163 Positive - C1D28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 4 | 5 | 5 | 3 | 0 | 0
  CD163 Positive - C1D28 |  |  |  |  |  |  |  |  |  |  | -4.1 [-21 to 1072] | -58.4 [-98 to -19] | 106.3 [-67 to 511] | -14.7 [-57 to 91] | 65.5 [-31 to 666] | 1.0 [-96 to 61] |  |
  CD163 Positive - C2D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 2
  CD163 Positive - C2D1 |  |  |  |  |  |  |  |  |  |  | -58.3 [-94 to -22] |  |  |  |  | -41.3 [-61 to -33] |  | 39.3 [-1 to 79]
  CD68 Positive - C0D7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD68 Positive - C0D7 |  |  |  |  |  |  | -70.2 [-91 to 107] | -17.1 [-64 to -2] |  |  |  |  |  |  |  |  |  |
  CD68 Positive - C0D14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD68 Positive - C0D14 |  |  |  |  |  |  | 57.7 [-12 to 128] | 7.9 [-8 to 24] |  |  |  |  |  |  |  |  |  |
  CD68 Positive - C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD68 Positive - C1D1 |  |  |  |  |  |  | 294.2 [203 to 385] | 17.8 [-39 to 102] |  |  |  |  |  |  |  |  |  |
  CD68 Positive - C1D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 2 | 0 | 0
  CD68 Positive - C1D15 |  |  |  |  |  |  | 2.9 [-26 to 185] | -26 [-26 to -26] |  |  |  | -4.0 [-27 to 58] | 81 [81 to 81] | 162.4 [150 to 175] |  | 92.5 [20 to 165] |  |
  CD68 Positive - C1D16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD68 Positive - C1D16 |  |  |  |  |  |  |  |  |  |  | 272 [272 to 272] |  |  |  |  |  |  |
  CD68 Positive - C1D28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 4 | 5 | 6 | 3 | 0 | 0
  CD68 Positive - C1D28 |  |  |  |  |  |  |  |  |  |  | 31.5 [-60 to 296] | -70.7 [-92 to -49] | 96.2 [-50 to 1106] | -38.3 [-88 to 121] | 96.2 [-25 to 179] | -4.3 [-46 to 102] |  |
  CD68 Positive - C2D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 1
  CD68 Positive - C2D1 |  |  |  |  |  |  |  |  |  |  | -26.9 [-50 to -4] |  |  |  |  | -40.0 [-54 to -33] |  | -66 [-66 to -66]

11. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) as determined by Investigator was defined as the number of participants with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) (per RECIST 1.1 criteria) divided by the number of all treated participants. Progression is defined as at least 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors. Complete response (CR)= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response (PR)= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose until disease progression, or the last response recorded (up to approximately 5 years)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 24
Percent of participants | 60.0 [26.2 to 87.8] | 25.0 [3.2 to 65.1] | 0 [0.0 to 30.8] | 18.2 [2.3 to 51.8] | 0 [0.0 to 36.9] | 0 [0.0 to 41.0] | 0 [0.0 to 41.0] | 0 [0.0 to 28.5] | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 9.4 [2.0 to 25.0] | 9.4 [2.0 to 25.0] | 19.2 [6.6 to 39.4] | 22.9 [10.4 to 40.1] | 17.1 [6.6 to 33.6] | 21.9 [9.3 to 40.0] | 0 [0.0 to 14.2] | 8.3 [1.0 to 27.0]

12. Primary Outcome: Duration of Response (DoR)
Description: Duration of Response (DOR), computed for all treated participants with a best overall response (BOR) of complete response (CR) or partial response (PR), is defined as the time between the date of first response (CR or PR) and the date of first documented disease progression as determined by RECIST 1.1 or death due to any cause, whichever occurs first, ie., DOR = disease progression date/death date -first response date + 1. For participants who remain alive and have not progressed, DOR will be censored on the date of their last tumor assessment.
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to date of disease progression or death, whichever occurs first (up to approximately 5 years)
Population: All treated participants who achieved complete or partial response and were not censored
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 6 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 7 | 6 | 7 | 0 | 2
Weeks | 159.00 [47.00 to NA] — Upper limit not calculated due to insufficient number of events | NA [16.43 to NA] — Median and upper limit not calculated due to insufficient number of events |  | NA [24.14 to NA] — Median and upper limit not calculated due to insufficient number of events |  |  |  |  |  |  | 74.14 [32.14 to NA] — Upper limit not calculated due to insufficient number of events | 56.57 [40.17 to NA] — Upper limit not calculated due to insufficient number of events | 36.21 [16.14 to NA] — Upper limit not calculated due to insufficient number of events | 32.14 [17.14 to 37.29] | 37.14 [14.14 to NA] — Upper limit not calculated due to insufficient number of events | 20.57 [14.29 to 31.00] |  | NA [41.00 to NA] — Median and upper limit not calculated due to insufficient number of events

13. Primary Outcome: Progression Free Survival (PFS) Rate at 24 Weeks
Description: PFS rate is defined as the proportion of participants who were progression free at Week 24. PFS is defined as the time from first dose to the date of first objectively documented disease progression or death due to any cause, whichever occurs first. Progression is defined at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm.
  Complete response (CR)= Disappearance of all target lesions. Pathological lymph nodes must have short axis reduction to < 10 mm. Partial response (PR)= At least 30% decrease in sum of diameters of target lesions.
  Participants who died w/o prior progression were considered progressed on death date. Those alive and not progressed were censored on the last tumor assessment date. Those who started subsequent therapy without reported progression were censored at last tumor assessment prior to subsequent therapy. Those without post-baseline tumor assessment and alive were censored at first dose.
Time Frame: From first dose up to Week 24
Population: All treated participants who were assessed for progression free survival at Week 24
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 7 | 4 | 5 | 6 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 14 | 13 | 17 | 21 | 13 | 0 | 3
Proportion of Participants | 0.778 [0.3648 to 0.9393] | NA [NA to NA] — Not calculated due to insufficient number of participants who reached threshold | 0.556 [0.2042 to 0.8045] | 0.800 [0.4087 to 0.9459] |  |  |  | NA [NA to NA] — Not calculated due to insufficient number of participants who reached threshold |  |  | 0.357 [0.1699 to 0.5490] | 0.536 [0.3372 to 0.6996] | 0.691 [0.4361 to 0.8478] | 0.535 [0.3512 to 0.6888] | 0.636 [0.4495 to 0.7746] | 0.467 [0.2779 to 0.6358] |  | NA [NA to NA] — Not calculated due to insufficient number of participants who reached threshold

14. Secondary Outcome: Maximim Concentration (Cmax)
Description: Cmax is defined as the maximum plasma concentration of the analytes at the prespecified timepoints.
Time Frame: From first dose up to the prespecified timepoints, C0D1, C0D14, and C2D1
Population: Pharmacokinetic evaluable participants - all participants who received at least one dose of medicine and have corresponding evaluable plasma or serum concentration data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 2 | 18 | 15 | 0 | 20 | 0 | 0 | 0 | 0
ng/mL
  C0D1 - BMS-813160: number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-813160 | 620.4 (250.60) | 2204.1 (961.90) | 828.4 (458.03) | 2419.0 (1203.53) | 486.3 (137.69) | 1896.3 (1421.89) | 1179.1 (605.50) | 276.28 (141.915) | 1580.0 (NA) — Standard deviation not calculated due to insufficient number of events | 807.0 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |
  C0D1 - BMS-939429: number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-939429 | 172.23 (103.837) | 435.6 (284.14) | 207.63 (142.559) | 545.7 (218.89) | 92.33 (50.015) | 539.1 (465.93) | 237.63 (188.286) | 54.82 (23.716) | 504.0 (NA) — Standard deviation not calculated due to insufficient number of events | 72.50 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |
  C0D14 - BMS-813160: number analyzed (Participants) | 8 | 4 | 7 | 5 | 6 | 2 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-813160 | 927.1 (513.88) | 4152.5 (2010.23) | 1060.3 (830.04) | 3274.0 (884.15) | 701.5 (284.59) | 1793.5 (1607.25) | 653.3 (298.08) | 80.00 (19.408) | 1370.0 (NA) — Standard deviation not calculated due to insufficient number of events | 1680.0 (961.67) |  |  |  |  |  |  |  |
  C0D14 - BMS-939429: number analyzed (Participants) | 8 | 4 | 7 | 5 | 6 | 2 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-939429 | 317.90 (290.209) | 658.3 (143.17) | 409.63 (382.471) | 792.2 (503.92) | 183.08 (190.050) | 326.0 (241.83) | 165.83 (92.914) | 25.307 (16.6021) | 498.0 (NA) — Standard deviation not calculated due to insufficient number of events | 265.40 (235.608) |  |  |  |  |  |  |  |
  C2D1 - BMS-813160: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 15 | 0 | 20 | 0 | 0 | 0 | 0
  C2D1 - BMS-813160 | 1153.1 (617.97) | 3280.0 (777.82) |  |  |  |  |  |  |  |  | 903.9 (578.56) | 357.55 (264.384) |  | 796.2 (472.48) |  |  |  |
  C2D1 - BMS-939429: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1 - BMS-939429 | 254.1 (140.73) | 571.0 (376.42) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

15. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: Tmax is defined as the time in hours of the maximum observed plasma concentration
Time Frame: From first dose up to the prespecified timpoints, C0D1, C0D14, AND C2D1
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 2 | 18 | 15 | 0 | 20 | 0 | 0 | 0 | 0
Hours
  C0D1 - BMS-813160: number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-813160 | 2.000 [0.50 to 4.00] | 0.500 [0.47 to 4.00] | 3.017 [2.00 to 4.02] | 2.492 [0.73 to 5.98] | 2.492 [0.52 to 11.92] | 2.983 [0.58 to 8.92] | 3.00 [0.50 to 6.00] | 1.992 [0.50 to 3.00] | 2.0 [2 to 2] | 3.950 [3.95 to 3.95] |  |  |  |  |  |  |  |
  C0D1 - BMS-939429: number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-939429 | 3.500 [0.50 to 6.25] | 1.000 [0.50 to 4.00] | 3.508 [1.00 to 11.98] | 3.000 [0.73 to 5.98] | 3.000 [1.0 to 11.92] | 2.083 [1.08 to 8.92] | 3.000 [1.00 to 6.00] | 2.000 [0.98 to 4.00] | 2.0 [2 to 2] | 1.950 [1.95 to 1.95] |  |  |  |  |  |  |  |
  C0D14 - BMS-813160: number analyzed (Participants) | 8 | 4 | 7 | 5 | 6 | 2 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-813160 | 3.000 [0.55 to 3.03] | 1.825 [0.50 to 3.00] | 2.917 [0.92 to 15.70] | 2.983 [0.50 to 4.00] | 2.875 [0.50 to 3.00] | 2.0 [1 to 3] | 2.000 [1.00 to 3.02] | 1.00 [0.5 to 4.0] | 2.02 [2.02 to 2.02] | 2.542 [2.00 to 3.08] |  |  |  |  |  |  |  |
  C0D14 - BMS-939429: number analyzed (Participants) | 8 | 4 | 7 | 5 | 6 | 2 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-939429 | 3.000 [0.98 to 4.00] | 1.825 [0.50 to 3.00] | 3.000 [1.08 to 15.70] | 2.983 [1.00 to 4.00] | 2.875 [1.17 to 3.00] | 2.492 [1.98 to 3.00] | 3.000 [1.00 to 4.02] | 1.0 [1 to 6] | 2.02 [2.02 to 2.02] | 3.117 [2.00 to 4.23] |  |  |  |  |  |  |  |
  C2D1 - BMS-813160: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 15 | 0 | 20 | 0 | 0 | 0 | 0
  C2D1 - BMS-813160 | 3.000 [0.98 to 4.23] | 1.000 [0.47 to 4.03] |  |  |  |  |  |  |  |  | 2.033 [0.50 to 14.10] | 2.067 [0.50 to 8.10] |  | 3.992 [0.50 to 16.17] |  |  |  |
  C2D1 - BMS-939429: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1 - BMS-939429 | 3.000 [2.00 to 4.23] | 1.000 [0.97 to 4.03] |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

16. Secondary Outcome: Trough Observed Plasma Concentration (Ctrough)
Description: Ctrough is defined as the concentration reached by a drug immediately before the next dose is administered
Time Frame: From first dose up to prespecified timepoints, C0D1, C5D1, C0D1, C1D15, C5D1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 6 | 3 | 4 | 4 | 5 | 1 | 2 | 2 | 1 | 2 | 11 | 16 | 3 | 7 | 6 | 0 | 1 | 1
ng/mL
  C0D1 - BMS-813160: number analyzed (Participants) | 6 | 3 | 4 | 4 | 5 | 1 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-813160 | 283.70 (207.784) | 84.30 (46.169) | 292.0 (154.31) | 74.05 (72.127) | 157.28 (92.311) | 137.0 (NA) — Standard deviation not calculated due to insufficient number of events | 57.10 (54.871) | 5.485 (2.4395) | 77.40 (NA) — Standard deviation not calculated due to insufficient number of events | 154.05 (139.936) |  |  |  |  |  |  |  |
  C5D1 - BMS-813160: number analyzed (Participants) | 6 | 3 | 4 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C5D1 - BMS-813160 | 268.80 (216.882) | 129.40 (89.944) | 176.0 (NA) — Standard deviation not calculated due to insufficient number of events | 15.30 (NA) — Standard deviation not calculated due to insufficient number of events | 323.0 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |  |  |  |  |  |
  C0D1 - BMS-939429: number analyzed (Participants) | 6 | 3 | 4 | 4 | 5 | 1 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-939429 | 172.63 (264.187) | 31.40 (10.689) | 180.88 (195.959) | 72.95 (55.542) | 47.60 (10.412) | 31.50 (NA) — Standard deviation not calculated due to insufficient number of events | 63.45 (60.175) | 4.950 (2.3052) | 90.30 (NA) — Standard deviation not calculated due to insufficient number of events | 71.65 (55.649) |  |  |  |  |  |  |  |
  C1D15 - BMS 939429: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 16 | 3 | 7 | 5 | 0 | 1 | 0
  C1D15 - BMS 939429 |  |  |  |  |  |  |  |  |  |  | 191.33 (84.266) | 24.106 (18.445) | 275.7 (164.34) | 116.04 (29.696) | 145.00 (99.293) |  | 283.0 (NA) — Standard deviation not calculated due to insufficient number of events |
  C5D1 - BMS-939429: number analyzed (Participants) | 6 | 3 | 4 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 11 | 12 | 1 | 5 | 6 | 0 | 0 | 1
  C5D1 - BMS-939429 | 55.78 (31.877) | 15.95 (4.172) | 155.0 (NA) — Standard deviation not calculated due to insufficient number of events | 10.50 (NA) — Standard deviation not calculated due to insufficient number of events | 65.20 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  | 186.21 (131.457) | 12.439 (6.9685) | 195.0 (NA) — Standard deviation not calculated due to insufficient number of events | 191.44 (113.725) | 222.65 (154.316) |  |  | 390.0 (NA) — Standard deviation not calculated due to insufficient number of events

17. Secondary Outcome: Area Under Curve (AUC) 0-8
Description: Area Under Curve (AUC) is defined as the area under the plot of plasma concentration of a drug versus time after dosage measured at 8 hours post-dose
Time Frame: From first dose up to prespecified timepoints- C0D1, C2D1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 8 | 7 | 7 | 6 | 1 | 1 | 9 | 13 | 0 | 14 | 0 | 0 | 1 | 0
ug*h/mL
  C0D1 - BMS-813160: number analyzed (Participants) | 10 | 7 | 9 | 10 | 8 | 6 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-813160 | 2300.018 (976.4608) | 7069.265 (2452.4213) | 2725.390 (1365.3562) | 7884.381 (3968.4940) | 1534.932 (518.2172) | 6593.904 (3603.5286) | 3533.737 (1931.7752) | 878.051 (535.3197) | 4440.313 (NA) — Standard deviation not calculated due to insufficient number of events | 3656.713 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |
  C0D1 - BMS-939429: number analyzed (Participants) | 9 | 7 | 9 | 10 | 8 | 6 | 7 | 6 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-939429 | 652.848 (363.5925) | 1783.336 (856.0103) | 936.394 (826.5807) | 2302.092 (1023.3978) | 342.534 (157.1350) | 2147.888 (1415.6386) | 942.398 (620.1018) | 210.938 (106.5352) | 1919.228 (NA) — Standard deviation not calculated due to insufficient number of events | 411.410 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |
  C2D1 - BMS-813160: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 13 | 0 | 14 | 0 | 0 | 0 | 0
  C2D1 - BMS-813160 | 5348.973 (2506.2558) | 11967.560 (4586.3823) |  |  |  |  |  |  |  |  | 4838.264 (2750.7756) | 1483.423 (1236.0374) |  | 3821.887 (2221.2474) |  |  |  |
  C2D1 - BMS-939429: number analyzed (Participants) | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1 - BMS-939429 | 1410.415 (837.4895) | 2403.182 (1144.3271) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

18. Secondary Outcome: Area Under Curve (AUC) 0-24
Description: as for outcome 17
Time Frame: From first dose up to prespecified timepoints-C0D1, C2D1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 0 | 7 | 0 | 9 | 0 | 5 | 7 | 6 | 0 | 1 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0
ug*h/mL
  C0D1 - BMS-813160: number analyzed (Participants) | 0 | 7 | 0 | 9 | 0 | 5 | 7 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-813160 |  | 9383.385 (2842.8397) |  | 11726.669 (6439.1376) |  | 10447.179 (2995.9347) | 4829.881 (2696.4668) | 1275.314 (799.8262) |  | 7687.658 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |
  C0D1 - BMS-939429: number analyzed (Participants) | 0 | 7 | 0 | 8 | 0 | 5 | 7 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-939429 |  | 2638.062 (977.2502) |  | 3991.522 (1636.3573) |  | 3905.941 (1852.8415) | 1660.159 (991.0121) | 341.0396 (160.4425) |  | 940.294 (NA) — Standard deviation not calculated due to insufficient number of events |  |  |  |  |  |  |  |
  C2D1 - BMS-813160: number analyzed (Participants) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1 - BMS-813160 |  | 17890.458 (9212.5646) |  |  |  |  |  |  |  |  |  | 2050.804 (997.6990) |  |  |  |  |  |
  C2D1 - BMS-939429: number analyzed (Participants) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C2D1 - BMS-939429 |  | 3958.779 (1632.3781) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

19. Secondary Outcome: Apparent Total Body Clearance (CLT/F)
Description: The total body clearance (CLT/F) is defined as the volume of plasma completely cleared of drug per unit time
Time Frame: From first dose up to prespecified timepoints-C0D1, C2D14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 8 | 5 | 7 | 4 | 6 | 2 | 3 | 2 | 1 | 2 | 9 | 13 | 0 | 10 | 0 | 0 | 0 | 0
mL/min
  C0D14 - BMS-813160: number analyzed (Participants) | 8 | 4 | 7 | 4 | 6 | 2 | 3 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-813160 | 1163.173 (588.1385) | 744.746 (361.5390) | 1521.863 (1277.8075) | 826.468 (300.1738) | 1602.009 (1123.8919) | 961.379 (235.4622) | 1688.813 (1022.7160) | 4950.110 (781.0155) | 1135.947 (NA) — Standard deviation not calculated due to insufficient number of events | 1032.434 (850.2203) |  |  |  |  |  |  |  |
  C2D1 - BMS-813160: number analyzed (Participants) | 6 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 13 | 0 | 10 | 0 | 0 | 0 | 0
  C2D1 - BMS-813160 | 956.446 (596.7553) | 683.958 (322.7045) |  |  |  |  |  |  |  |  | 1115.087 (851.2513) | 1813.987 (1920.2627) |  | 1440.516 (733.5156) |  |  |  |

20. Secondary Outcome: Renal Clearance (CLR)
Description: Renal clearance is defined as the rate at which the analytes were removed from the plasma by the kidneys.
Time Frame: From first dose up to prespecified timepoints-C0D1, C0D14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 7 | 4 | 6 | 3 | 7 | 3 | 5 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
mL/min
  C0D1 - BMS-813160: number analyzed (Participants) | 7 | 4 | 6 | 3 | 7 | 3 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-813160 | 212.411 (191.8961) | 275.309 (277.2659) | 139.012 (107.2006) | 165.327 (77.8766) | 155.820 (119.3858) | 181.930 (9.1130) | 248.003 (82.6974) | 236.781 (62.8689) |  |  |  |  |  |  |  |  |  |
  C0D1 - BMS-939429: number analyzed (Participants) | 6 | 4 | 6 | 3 | 7 | 3 | 5 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D1 - BMS-939429 | 74.298 (44.8889) | 175.109 (187.5683) | 68.184 (52.1580) | 77.744 (34.8177) | 81.027 (65.1050) | 98.733 (6.2562) | 140.597 (41.7347) | 128.943 (26.7782) |  | 62.007 |  |  |  |  |  |  |  |
  C0D14 - BMS-813160: number analyzed (Participants) | 7 | 2 | 4 | 2 | 4 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-813160 | 185.926 (56.5866) | 124.400 (52.1454) | 260.786 (120.8954) | 168.274 (72.7581) | 158.238 (82.5905) | 194.009 (50.1111) | 283.842 (109.4518) | 149.271 (72.0204) |  | 115.147 |  |  |  |  |  |  |  |
  C0D14 - BMS-939429: number analyzed (Participants) | 7 | 2 | 3 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C0D14 - BMS-939429 | 101.042 (27.5043) | 76.285 (30.5071) | 145.662 (73.3215) | 91.490 (43.8006) | 87.068 (43.9667) | 111.649 (32.4552) |  |  |  |  |  |  |  |  |  |  |  |

21. Secondary Outcome: Number of Participants Who Were Anti-Drug Antibody (ADA) Positive
Description: The number of participants who are anti-drug antibody positive. ADA-positive participant is a participant with at least 1 ADA-positive sample relative to baseline after initiation of the treatment. ADA-positive sample is in a participant who is baseline ADA negative or with an ADA titer to be at least 4-fold or greater than baseline positive titer.
Time Frame: From first dose up to prespecified timepoints-C1D1, C1D15, C2D1, C3D1, C5D1, C9D1
Population: All treated participants with baseline measurements and at least one positive ADA assessment of Nivolumab
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIRI | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
Number analyzed (Participants) | 10 | 8 | 10 | 11 | 8 | 7 | 7 | 11 | 1 | 2 | 32 | 32 | 26 | 35 | 35 | 32 | 24 | 33
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 5.5 years). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 3 years).
Description: The 9 crossover participants are counted in the arm in which they experienced the adverse event.
Groups:
- Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIR: First-line treatment BMS-813160 300 mg twice a day in combination with FOLFIRI in participants with metastatic colorectal cancer
- Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI: Second-line treatment FOLFIRI in participants with colorectal cancer.
Arm/Group | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIR | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO
All-Cause Mortality (participants affected / at risk) | 6/10 | 6/8 | 8/10 | 8/11 | 6/8 | 6/7 | 6/7 | 7/11 | 1/1 | 2/2 | 26/32 | 28/32 | 17/26 | 33/35 | 34/35 | 26/32 | 20/24 | 25/33
Serious Adverse Events (participants affected / at risk) | 5/10 | 5/8 | 5/10 | 7/11 | 5/8 | 6/7 | 6/7 | 6/11 | 1/1 | 2/2 | 12/32 | 12/32 | 6/26 | 24/35 | 22/35 | 15/32 | 17/24 | 19/33
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8 | 9/10 | 11/11 | 8/8 | 7/7 | 7/7 | 10/11 | 1/1 | 2/2 | 32/32 | 31/32 | 25/26 | 35/35 | 34/35 | 31/32 | 19/24 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIR (N=10) | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI (N=8) | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB (N=10) | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB (N=11) | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO (N=8) | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO (N=7) | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO (N=7) | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO (N=11) | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO (N=1) | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO (N=2) | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI (N=32) | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI (N=32) | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI (N=26) | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB (N=35) | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO (N=35) | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB (N=32) | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO (N=24) | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 3 | 2 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cholangitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fournier's gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis sapovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 2 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Splenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wrong product administered (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 7 | 8
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1-Arm A-Cohort 1: 1L CRC/BMS300BID + FOLFIR (N=10) | Part 1-Arm A-Cohort 2: 1L CRC/BMS600QD + FOLFIRI (N=8) | Part 1-Arm B-Cohort 1: 1L PC/BMS300BID + GEM/NAB (N=10) | Part 1-Arm B-Cohort 2: 1L PC/BMS600QD + GEM/NAB (N=11) | Part 1-Arm C-Cohort 1: 2/3L CRC MSS/BMS300BID + NIVO (N=8) | Part 1-Arm C-Cohort 2: 2/3L CRC MSS/BMS600QD + NIVO (N=7) | Part 1-Arm C-Cohort 3: 2/3L CRC MSS/BMS300QD + NIVO (N=7) | Part 1-Arm C-Cohort 4: 2/3L CRC MSS/BMS150QD + NIVO (N=11) | Part 1-Arm C-Cohort 5: 2L PC/BMS300BID + NIVO (N=1) | Part 1-Arm C-Cohort 6: 2L PC/BMS600QD + NIVO (N=2) | Part 2-Arm A-Cohort 1a: 2L CRC/BMS300BID + FOLFIRI (N=32) | Part 2-Arm A-Cohort 1b: 2L CRC/BMS150QD + FOLFIRI (N=32) | Part 2-Arm A-Cohort 1C: 2L CRC/FOLFIRI (N=26) | Part 2-Arm B-Cohort 3a: 1L PC/BMS300BID + GEM/NAB (N=35) | Part 2-Arm B-Cohort 3b: 1L PC/BMS300BID + GEM/NAB + NIVO (N=35) | Part 2-Arm B-Cohort 3C: 1L PC/GEM/NAB (N=32) | Part 2-Arm C-Cohort 4: 2L PC/BMS300BID + NIVO (N=24) | Part 2-Arm C-Cohort 5: 2/3L CRC MSS /BMS300BID + NIVO (N=33)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 5 | 5 | 4 | 3 | 2 | 1 | 0 | 0 | 5 | 5 | 5 | 21 | 20 | 20 | 7 | 6
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 4 | 4 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 7 | 8 | 7 | 7 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 9 | 12 | 6 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5 | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 2 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 0 | 0 | 3 | 2 | 0 | 0 | 10 | 6 | 3 | 13 | 9 | 8 | 5 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 1 | 3 | 3 | 2 | 3 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal rash (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4 | 5 | 3 | 1 | 1 | 3 | 3 | 0 | 1 | 13 | 7 | 8 | 16 | 15 | 12 | 4 | 2
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 3 | 2 | 3 | 1 | 3 | 3 | 1 | 0 | 13 | 14 | 15 | 15 | 19 | 13 | 6 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 6 | 2 | 1 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 2 | 4 | 3 | 1 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 3 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 6 | 4 | 7 | 2 | 1 | 4 | 2 | 0 | 1 | 12 | 12 | 12 | 23 | 21 | 14 | 9 | 6
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 7 | 5 | 7 | 7 | 6 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4 | 3 | 1 | 1 | 5 | 2 | 1 | 1 | 6 | 10 | 8 | 10 | 11 | 9 | 5 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 5 | 3 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 6 | 5 | 3 | 1 | 1
Cyst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 7 | 5 | 5 | 3 | 3 | 4 | 0 | 1 | 13 | 11 | 15 | 23 | 27 | 19 | 10 | 9
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 4 | 1 | 3 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 2 | 2 | 0 | 1 | 1
Oedema peripheral (General disorders) | 2 | 0 | 1 | 5 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 15 | 12 | 11 | 2 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 2 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 3 | 0 | 0 | 5 | 4 | 1 | 11 | 15 | 10 | 5 | 6
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 1 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 0
Pyuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 3 | 1 | 2 | 3 | 2 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 3 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular access site rash (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 3 | 4 | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 10 | 10 | 10 | 3 | 2
Amylase increased (Investigations) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 3 | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 3 | 2 | 2 | 0 | 1 | 3 | 0 | 0 | 2 | 1 | 2 | 8 | 8 | 9 | 3 | 7
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 2 | 3 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 4 | 0 | 9 | 10 | 9 | 7 | 5
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 2 | 4 | 5 | 2
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 3 | 0
Lipase increased (Investigations) | 4 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 6 | 1 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 3 | 4 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 14 | 8 | 8 | 7 | 10 | 15 | 0 | 1
Platelet count decreased (Investigations) | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 8 | 7 | 9 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 3 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 3 | 2 | 2 | 7 | 9 | 5 | 5 | 5
White blood cell count decreased (Investigations) | 2 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 9 | 8 | 6 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 2 | 5 | 4 | 2 | 2 | 1 | 0 | 0 | 10 | 6 | 4 | 17 | 16 | 12 | 7 | 10
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 5 | 2 | 3 | 1 | 1 | 3 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 9 | 5 | 5 | 7 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 2 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 10 | 8 | 6 | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 7 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 1 | 4 | 6 | 7 | 4 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 4 | 4 | 4 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 8 | 7 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 5 | 5 | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 6 | 6 | 5 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 5 | 3 | 8 | 3 | 2 | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 4 | 1 | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 2 | 4 | 2 | 2 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 9 | 6 | 7 | 0 | 4
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 2 | 2 | 8 | 5 | 5 | 1 | 1
Headache (Nervous system disorders) | 1 | 3 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 4 | 9 | 3 | 0 | 3
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Narcolepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 6 | 6 | 5 | 3 | 3
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 17 | 11 | 8 | 4 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 3 | 0 | 1 | 4
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 4 | 3 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 4 | 1 | 1 | 3 | 5
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 0 | 0 | 3 | 4 | 3 | 11 | 11 | 3 | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 3 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 10 | 9 | 6 | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 4 | 4 | 4 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 3 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 4 | 13 | 11 | 12 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 3 | 5 | 3 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 9 | 13 | 3 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 8 | 4 | 0 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 2 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 4 | 3 | 4 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 3 | 4 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03184870/Prot_SAP_000.pdf